

# NON-INTERVENTIONAL STATISTICAL ANALYSIS PLAN FOR SECONDARY DATA COLLECTION STUDY

# **VERSION HISTORY**

| Version | Effective Date | Change Type<br>(New, Revise,<br>Admin) | Summary of Revisions |
|---|---|---|---|
| 1.0 | 22-May-2023 | New | - |



# Non-Interventional Study Protocol < B9991052>

A Multicenter, Non-Interventional, Retrospective, Observational Study Evaluating Real-World Treatment Outcomes in Japanese Patients with Metastatic Renal Cell Carcinoma (mRCC) Treated using Avelumab plus Axitinib as First-line Therapy: J-DART2

Statistical Analysis Plan (SAP)

Version: 1.0

Author: PPD

Date: 22-May-2023

# **TABLE OF CONTENTS**

| 1 | $\mathbf{A}\mathbf{N}$ | IENDMENTS FROM PREVIOUS VERSION(S) | 5 |
|---|---|---|---|
| 2 | INT | TRODUCTION | 5 |
| | 2.1 | STUDY DESIGN | 5 |
| | Stu | dy population | |
| | | 'a source | |
| | | atment/cohort labels | |
| | 2.2 | STUDY OBJECTIVES | |
| 3 | HY | POTHESES AND DECISION RULES | 6 |
| | 3.1 | STATISTICAL HYPOTHESES | 6 |
| | 3.2 | STATISTICAL DECISION RULES | 6 |
| 4 | AN | ALYSIS SETS/POPULATIONS | 6 |
| | 4.1 | FULL ANALYSIS SET (FAS) | 6 |
| | 4.2 | SAFETY ANALYSIS SET | |
| | 4.3 | OTHER ANALYSIS SET | |
| | 4.4 | SUBGROUPS | 7 |
| 5 | EN | DPOINTS AND COVARIATES | 7 |
| | 5.1 | EFFICACY/EFFECTIVENESS ENDPOINT(S) | 7 |
| | 5.2 | SAFETY ENDPOINTS | . 10 |
| | <b>CC</b> 5.4 | | |
| | | Covariates | |
| 6 | HA | NDLING OF MISSING VALUES | . 16 |
| 7 | ST | ATISTICAL METHODOLOGY AND STATISTICAL ANALYSES | . 16 |
| | 7.1 | STATISTICAL METHODS | . 16 |
| | 7.2 | STATISTICAL ANALYSES | |
| | 7.2. | | . 17 |
| | 7.2. | 2 Analysis of primary, secondary, and CCI | . 17 |
| | | .2.2.1 Demographic and clinical characteristics of patients | |
| | | 2.2.3 Overall survival (OS) | |
| | | 2.2.4 Objective response rate (ORR) | |
| | | .2.2.5 Best overall response for primary lesions | |
| | | .2.2.6 Time to treatment discontinuation (TTD) of avelumab plus axitinib | |
| | | ombination therapy as first-line therapy | . 22 |
| | | .2.2.7 Treatment patterns for avelumab plus axitinib combination therapy as | |
| | f | irst-line therapy in a real-world setting | . 23 |

7.2.2.8 Clinical use of corticosteroids for immune-related adverse events (irAEs) occurring during the course of avelumab plus axitinib combination 7.2.2.9 Pre-treatment and treatment of infusion-related reactions caused by 7.2.2.10 Subsequent treatment of avelumab plus axitinib combination therapy 8 9 APPENDIXES 30 *A1.2 Further definition of endpoints.* APPENDIX 2: ADDITIONAL STATISTICAL METHODOLOGY DETAILS ... 30 10.2 APPENDIX 3: DIAGNOSIS AND PROCEDURE CODES USED IN THE STUDY ........ 30

#### 1 AMENDMENTS FROM PREVIOUS VERSION(S)

Not applicable

#### 2 INTRODUCTION

#### 2.1 STUDY DESIGN

The present study is a multicenter, non-interventional, retrospective, medical chart review of patients with metastatic renal cell carcinoma (mRCC) who received avelumab plus axitinib as first-line therapy in Japan between December 20, 2019, and October 17, 2022.

The source population comprised patients who initiated avelumab plus axitinib as first-line therapy between December 20, 2019, and October 17, 2022.

### **Study population**

This retrospective chart review will evaluate patient data derived from the existing medical records of all enrolled patients. All decisions regarding the clinical management and treatment of the patients are made by the investigator as part of standard care in a real-world setting and are not contingent upon the patient's participation in the study. Data will be collected at each study site (if available).

The study period will range from December 20, 2019, to October 31, 2022. Patients with an index date between December 20, 2019, and October 17, 2022, will be enrolled in this study. To ensure a two-week follow-up period, patients with an index date between December 20, 2019, and October 17, 2022, will be included. The two-week follow-up period is determined based on the dosing interval for avelumab, considering that the time of initiation of avelumab and axitinib may differ.

Index date: The date of the first prescription of avelumab plus axitinib combination therapy.

Observation period: Patients will be followed-up from the index date to October 31, 2022.

\*The date of the first prescription of avelumab plus axitinib combination therapy is the administration start date of the drug initiated first.

#### **Data source**

Considering the retrospective nature of the study, all data will be collected from patient medical records at the participating study sites.

#### Treatment/cohort labels

Avelumab plus axitinib combination therapy

#### 2.2 STUDY OBJECTIVES

*Primary objective* 

To describe the demographic and clinical characteristics of Japanese patients with mRCC treated using avelumab plus axitinib as a first-line therapy in a real-world setting.

# Secondary objectives

- To evaluate the treatment outcomes of avelumab plus axitinib as first-line therapy for patients with mRCC in a real-world setting, as determined by the following endpoints:
  - Real-world progression-free survival (PFS).
  - Overall survival (OS).
  - *Objective response rate (ORR).*
  - Best overall response (BOR) for primary lesions.
  - Time to treatment discontinuation (TTD) of avelumab plus axitinib as first-line therapy.
- To describe the treatment patterns for avelumab plus axitinib as first-line therapy in a real-world setting.
- To describe the clinical applicability of corticosteroids for immune-related adverse events (irAEs) occurring during the course of avelumab plus axitinib combination therapy.
- To describe the pre-treatment and treatment of infusion-related reactions caused by avelumab.
- To describe the subsequent treatment of avelumab plus axitinib combination therapy.



#### 3 HYPOTHESES AND DECISION RULES

#### 3.1 STATISTICAL HYPOTHESES

This study is not intended to test hypotheses.

#### 3.2 STATISTICAL DECISION RULES

A two-sided 95% confidence interval will be calculated for interval estimation. In addition, no multiplicity adjustment will be performed.

#### 4 ANALYSIS SETS/POPULATIONS

#### 4.1 FULL ANALYSIS SET (FAS)

The FAS will comprise patients who meet the inclusion criteria and do not meet the exclusion criteria.

#### **Inclusion criteria**

1) Diagnoses of mRCC based on the General Rule for Clinical and Pathological Studies on RCC (Fifth Edition) before the administration of avelumab plus axitinib

as first-line therapy. Patients with mRCC presenting with unresectable disease, either a unresectable locally advanced or metastatic disease.

- 2) Age over 18 years at the time of the first administering of avelumab plus axitinib a as first-line therapy for mRCC (baseline).
- 3) Index date from December 20, 2019, to October 17, 2022.

#### **Exclusion criteria**

- 1) Patients participating in a prospective interventional clinical trial assessing an investigational product during the observational period.
- 2) Patients (or a patient's legal representative) refusing to provide patient data during the consent process.

#### 4.2 SAFETY ANALYSIS SET

Not applicable

#### 4.3 OTHER ANALYSIS SET

Efficacy analysis set

The efficacy analysis set is a subset of the FAS comprising patients whose index date is prior to April 30, 2022, to ensure a 6-month follow-up period.

#### 4.4 SUBGROUPS

A subgroup analysis will be considered, including but not limited to the subgroups categorized by IMDC (International Metastatic RCC Database Consortium) risk group, age ( $\geq 75$  years or < 75 years), and the administration of corticosteroid therapy for irAE in the medical record.

#### 5 ENDPOINTS AND COVARIATES

Handling of data on the number of days

The number of days from the start date to the target date will be calculated as follows:

- The target date is earlier than the start date = Target date Start date
- The target date is on or after the start date = Target date Start date + 1

The number of days will be handled as follows:

 $\sqrt{1}$  week = 7 days

 $\sqrt{1}$  month = 30.4375 days

 $\sqrt{1 \text{ year}} = 365.25 \text{ days}$ 

In addition, missing data will be imputed with reference to "6. HANDLING OF MISSING VALUES."

#### 5.1 EFFICACY/EFFECTIVENESS ENDPOINT(S)

< Derivation of time-to-event variables >

| Item | Derivation method |
|---|---|
| Real-world progression-free survival (PFS) | Defined as the period from the start date of |
| | avelumab plus axitinib combination therapy to |

| | the date of first disease progression (clinical |
|---|---|
| | evaluation based on radiographic, clinical, and |
| | pathological examinations, as well as other |
| | evaluations by the principal investigator or co- |
| | investigator) or death from any cause, whichever |
| | occurs earlier. If there is no clinical record of |
| | death or disease progression, the following dates |
| | will be used for censoring, based on medical |
| | records: |
| | (1) If first-line therapy is ongoing, the final |
| | progression-free confirmation date or the date of |
| | the last hospital visit, whichever is earlier, will |
| | be used for censoring. |
| | (2) If second-line therapy has not been initiated |
| | after the end of first-line therapy, the final |
| | progression-free confirmation date or the date of |
| | the last hospital visit, whichever is earlier, will |
| | be used for censoring. |
| | (3) If second-line therapy has been initiated, the |
| | date of initiating the second-line therapy will be |
| | used for censoring. |
| | (4) If nephrectomy has been performed, the date |
| Reasons for real-world PFS events | of nephrectomy will be used for censoring. Reasons for real-world PFS events are defined as |
| Reasons for fear-world FFS events | follows: |
| | "Disease progression after the initiation of |
| | avelumab plus axitinib combination therapy" |
| | will be selected if there was disease progression |
| | after starting avelumab plus axitinib combination |
| | therapy. |
| | "Death" will be selected if the patient has died. |
| Reasons for censoring real-world PFS | Reasons for censoring real-world PFS are |
| | defined as follows: |
| | "No disease progression during or after first-line |
| | therapy" will be selected if first-line therapy is |
| | ongoing or if second-line therapy has not been |
| | initiated after the end of first-line therapy. |
| | "Second-line therapy started" will be selected if |
| | second-line therapy has been initiated. |
| | "Nephrectomy performed" will be selected if |
| | nephrectomy has been performed. |
| Overall survival (OS) | Defined as the period from the initiation of |
| | avelumab plus axitinib combination therapy to |
| | the date of death from any cause. If there is no |

| | record of death, the date when the survival of the |
|---|---|
| | patient was last confirmed on record (date of last |
| | hospital visit) will be used for censoring. |
| Time to treatment discontinuation (TTD) of | Defined as the period from the date of initiation |
| avelumab plus axitinib combination | of avelumab plus axitinib combination therapy to |
| therapy as first-line therapy | the date of ending treatment* for any reason |
| therapy as mist-fine therapy | (excluding discontinuation due to efficacy). |
| | In the case of discontinuation due to efficacy, |
| | the date of last administration will be used for |
| | censoring. If treatment has not ended, the date of |
| | the last hospital visit will be used for censoring. |
| | * The end date of treatment is the date of last |
| | avelumab administration + 13 days or the date of |
| | last axitinib administration, whichever occurs |
| | later, or the data-cut date, if performed earlier. |
| TTD of avelumab as first-line therapy | Defined as the period from the date of initiation |
| 112 of averaginae as first line alorapy | of avelumab to the date of ending |
| | administration* for any reason (excluding |
| | discontinuation due to efficacy). In the case of |
| | discontinuation due to efficacy, the date of the |
| | last avelumab administration will be used for |
| | censoring. |
| | If treatment has not ended, the date of the last |
| | hospital visit will be used for censoring. |
| | * The end date of avelumab therapy is the date of |
| | the last avelumab administration + 13 days or the |
| | data-cut date, whichever occurs earlier. |
| TTD of axitinib as first-line therapy | Defined as the period from the date of initiation |
| | of axitinib to the date of ending administration* |
| | for any reason (excluding discontinuation due to |
| | efficacy). In the case of discontinuation due to |
| | efficacy, the date of the last axitinib |
| | administration will be used for censoring. |
| | If treatment has not ended, the date of the last |
| | hospital visit will be used for censoring. |
| | * The end date of axitinib is the date of the last |
| D 0 1 TITE | axitinib administration. |
| Reasons for the TTD event | Reasons for TTD event are defined as follows: |
| | Disease progression/adverse event/other |
| Decree for consoning TTD | (death)/other (excluding death) |
| Reasons for censoring TTD | Reasons for censoring TTD are defined as |
| | follows: |
| | "Treatment ongoing" will be selected if the |
| | treatment is ongoing. |

| " discontinuation due to efficacy " will be selected in case of discontinuation due to |
|---|
| efficacy. |

# < Derivation of categorical variables >

| Item | Derivation method |
|---|---|
| Objective response to avelumab plus | Determination of the best overall response |
| axitinib combination therapy | (tumor assessment) is categorized as follow: |
| | "Objective response" when "CR" or "PR." |
| | "Non-objective response" when "SD," "PD," or |
| | "NE". |
| Objective response of primary lesions | Determination of the best overall response |
| | (tumor assessment) is categorized as follow: |
| | "Objective response" when "CR" or "PR." |
| | "Non-Objective response " when "SD," "PD," or |
| | "NE." |

CR, complete response; PR, partial response; PD, progressive disease; NE, not evaluable for response; SD, stable disease.

# **5.2 SAFETY ENDPOINTS**

Not applicable



PFIZER CONFIDENTIAL
CT24-WI-GL03-RF03 2.0 Non-Interventional Statistical Analysis Plan For Secondary Data Collection
Study 01-Jun-2020




# < Derivation of categorical variables >

| Item | Derivation method |
|---|---|
| Age (2 categories ) | Age is divided into the following categories: <75 years; ≥75 years |
| Age (3 categories ) | Age is divided into the following categories: <65 years; ≥65 years and <75 years; ≥75 years |
| Body mass index (BMI) (3 categories ) | BMI is divided into the following categories: <25 kg/m²; ≥25 kg/m²; Unknown |
| C-reactive protein (CRP) (3 categories ) | CRP is divided into the following categories: <5 mg/L; ≥5 mg/L; Unknown **Categorized as "Unknown" if CRP is missing (Not measured) |
| Estimated glomerular filtration rate (eGFR) (3 categories ) | eGFR is divided into the following categories:<br><60; ≥60; Unknown<br>※Categorized as "Unknown" if eGFR is missing<br>(Not measured) |
| Fuhrman grade (3 categories ) | Fuhrman grade is divided into the following categories: Grade 1 or Grade 2; Grade 3 or Grade 4; Unknown |

| No. 1 of the T | HXZ H '11 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 |
|---|---|
| Metastatic site: Lung | "Yes" will be selected if the presence or absence |
| | of metastasis is "Yes" and the metastatic site is |
| | "Lung." |
| | "No" will be selected if the presence or absence |
| | of metastasis is "Yes" and the metastatic site is |
| | not "Lung" or if the presence or absence of |
| | metastasis is "No." |
| | "Unknown" will be selected if the presence or |
| | absence of metastasis is "Unknown." |
| Metastatic site: Liver | "Yes" will be selected if the presence or absence |
| | of metastasis is "Yes" and the metastatic site is |
| | "Liver." |
| | "No" will be selected if the presence or absence |
| | of metastasis is "Yes" and the metastatic site is |
| | not "Liver" or if the presence or absence of |
| | metastasis is "No." |
| | "Unknown" will be selected if the presence or |
| | absence of metastasis is "Unknown." |
| Metastatic site: Bone | "Yes" will be selected if the presence or absence |
| | of metastasis is "Yes" and the metastatic site is |
| | "Bone." |
| | "No" will be selected if the presence or absence |
| | of metastasis is "Yes" and the metastatic site is |
| | not "Bone" or if the presence or absence of |
| | metastasis is "No." |
| | "Unknown" will be selected if the presence or |
| | absence of metastasis is "Unknown." |
| Metastatic site: Brain | "Yes" will be selected if the presence or absence |
| | of metastasis is "Yes" and the metastatic site is |
| | "Brain." |
| | "No" will be selected if the presence or absence |
| | of metastasis is "Yes" and the metastatic site is |
| | not "Brain" or if the presence or absence of |
| | metastasis is "No." |
| | "Unknown" will be selected if the presence or |
| | absence of metastasis is "Unknown." |
| Metastatic site: Regional lymph node | "Yes" will be selected if the presence or absence |
| | of metastasis is "Yes" and the metastatic site is |
| | "Regional lymph node." |
| | "No" will be selected if the presence or absence |
| | of metastasis is "Yes" and the metastatic site is |
| | absence of metastasis is "No." |
| | "No" will be selected if the presence or absence of metastasis is "Yes" and the metastatic site is not "Regional lymph node" or if the presence or |

| | "Unknown" will be selected if the presence or |
|---|---|
| | absence of metastasis is "Unknown." |
| Metastatic site: Distant lymph node | "Yes" will be selected if the presence or absence |
| | of metastasis is "Yes" and the metastatic site is a |
| | "Distant lymph node." "No" will be selected if |
| | the presence or absence of metastasis is "Yes" |
| | and the metastatic site is not a "Distant lymph |
| | node" or if the presence or absence of metastasis |
| | is "No." |
| | "Unknown" will be selected if the presence or |
| | absence of metastasis is "Unknown." |
| Metastatic site: Other | "Yes" will be selected if the presence or absence |
| | of metastasis is "Yes" and the metastatic site is |
| | "Other." |
| | "No" will be selected if the presence or absence |
| | of metastasis is "Yes" and the metastatic site is |
| | not "Other" or if the presence or absence of |
| | metastasis is "No." |
| | "Unknown" will be selected if the presence or |
| | absence of metastasis is "Unknown." |
| ECOG Performance Status (1) | ECOG Performance Status is divided into the |
| | following categories: |
| | 0; 1; ≥2 |
| ECOG Performance Status 2 | ECOG Performance Status is divided into the |
| | following categories: |
| | 0 or 1; $\geq$ 2 |
| Number of risk factors (7 categories) | The number of risk factors is divided into the |
| | following categories: |
| | 0; 1; 2; 3; 4; 5; 6 |
| Initial dose of avelumab [daily dose (mg)] | The initial dose of avelumab is divided into the |
| | following categories: |
| | <10 mg/kg; 10 mg/kg; >10 mg/kg |
| Initial dose of axitinib [daily dose (mg)] | The initial dose of axitinib is divided into the |
| | following categories: |
| | $<2 \text{ mg}; \ge 2 \text{ mg and } <5 \text{ mg}; \ge 5 \text{ mg and } <10 \text{ mg};$ |
| | <10 mg; 10 mg; >10 mg |
| Presence or absence of changes in the | "Yes" will be selected if the dose of avelumab |
| avelumab dose | was changed even once. |
| | "No" will be selected if the dose was unchanged. |
| Presence or absence of changes in the | "Yes" will be selected if the dose of avelumab |
| avelumab dose (dose reduction) | was changed (dose reduction) even once. |
| | "No" will be selected if the dose was unchanged |
| | (dose reduction). |

| Presence or absence of change in the dose | "Yes" will be selected if the dose of avelumab |
|---|---|
| of avelumab (dose increase) | was changed (dose increase) even once. |
| | "No" will be selected if the dose was unchanged. |
| Presence or absence of changes in the | "Yes" will be selected if the dose of axitinib was |
| axitinib dose | changed even once. |
| | "No" will be selected if the dose was unchanged. |
| Presence or absence of changes in the | "Yes" will be selected if the dose of axitinib was |
| axitinib dose (dose reduction) | changed (dose reduction) even once. |
| | "No" will be selected if the dose was unchanged. |
| Presence or absence of changes in the | "Yes" will be selected if the dose of axitinib was |
| axitinib dose (dose increase) | changed (dose increase) even once. |
| | "No" will be selected if the dose was unchanged. |
| Administration of high-dose corticosteroid | "Yes" will be selected if the prednisolone- |
| therapy for iRAE | equivalent* daily dose was ≥40 mg. |
| | Otherwise, "No" will be selected. |

\*In addition, the corticosteroid-equivalent dose (prednisolone-equivalent) is calculated as the dose of the drug × prednisolone conversion ratio, according to the table below:

| General name | Corresponding dose | Prednisolone |
|--------------------|--------------------|------------------|
| | (mg) | conversion ratio |
| Cortisone | 25 | 0.2 |
| Hydrocortisone | 20 | 0.25 |
| Prednisolone | 5 | 1 |
| Methylprednisolone | 4 | 1.25 |
| Triamcinolone | 4 | 1.25 |
| Dexamethasone | Approximately 0.75 | 6.67 |
| Betamethasone | Approximately 0.75 | 6.67 |

#### 5.4 COVARIATES

- Age (2 categories)
- Body mass index (BMI) (3 categories)
- C-reactive protein (CRP) (3 categories)
- Estimated glomerular filtration rate (eGFR) (3 categories)
- · Smoking history
- ECOG Performance Status
- ECOG Performance Status (1)
- ECOG Performance Status (2)
- Tumor histological type
- Presence or absence of sarcomatoid component
- Fuhrman grade (3 categories)
- Performance of nephrectomy
- · Metastatic site: Lung

Metastatic site: LiverMetastatic site: BoneMetastatic site: Brain

• Metastatic site: Regional lymph node

• Metastatic site: Distant lymph node

· Metastatic site: Other

• Number of metastatic organs (5 categories)

- Presence or absence of clinically important comorbidities
- Presence or absence of clinically important concomitant drugs
- Less than 1 year from diagnosis to the initiation of systemic therapy
- Karnofsky Performance Status <80%
- Hemoglobin value below the lower normal limit
- Corrected calcium value above the upper normal limit
- Neutrophil count above the upper normal limit
- Platelet count above the upper normal limit
- IMDC risk group
- Administration of corticosteroid therapy for irAEs

#### 6 HANDLING OF MISSING VALUES

An absence of data for analysis will be treated as missing values, and no special imputation processing will be performed using statistical methods. In addition, the missing data regarding dates will be treated as follows:

✓If "year" is unknown: Missing
✓If "month" is unknown: July
✓If "day" is unknown: day 15
✓If "month" and "day" are unknown: July 1

Other than the above, the imputation of the missing values will not be performed, unless otherwise specified.

If the above imputation measures result in the reversal of dates when calculating the number of days (e.g., the number of days from the initiation to the end of the treatment), it will not be adopted for analysis.

# 7 STATISTICAL METHODOLOGY AND STATISTICAL ANALYSES 7.1 STATISTICAL METHODS

#### Summary statistics

For summary statistics described in this plan, the following values will be calculated, unless otherwise specified:

Number of cases, number of missing cases, mean, standard deviation, minimum, quartiles, and maximum

#### Number of digits

The percentage (%) of frequency distribution will be rounded to one decimal place, unless otherwise specified, in the individual analysis items. Considering the summary statistics items (number of cases, number of missing cases, mean, standard deviation, minimum, quartiles, and maximum), mean, standard deviation, and quartiles will be rounded such that the decimal places are one digit lower than the original data.

#### 7.2 STATISTICAL ANALYSES

#### 7.2.1 Safety analyses

Not applicable

# 7.2.2 Analysis of primary, secondary, and

### **Analysis of primary endpoints**

# 7.2.2.1 Demographic and clinical characteristics of patients

Source: FAS, Efficacy analysis set

population

Endpoints : Continuous variables

Age Height Body weight

BMI

CRP eGFR

Number of metastatic organs

Number of risk factors

Observation duration (months)

#### Categorical variables

Age (2 categories)

Age (3 categories)

BMI (3 categories)

Gender

CRP (3 categories) eGFR (3 categories) Smoking history

ECOG Performance Status ECOG Performance Status (1)

ECOG Performance Status 2

Invasion depth (T factor)

Lymph node metastasis (N factor)

Distant metastasis (M factor)

Tumor histological type

Presence or absence of sarcomatoid component

Fuhrman grade

Fuhrman grade (3 categories)

Proteinuria

Performance of nephrectomy

Presence or absence of metastasis

Metastatic site

Metastatic site: Lung Metastatic site: Liver Metastatic site: Bone Metastatic site: Brain

Metastatic site: Regional lymph node Metastatic site: Distant lymph node

Metastatic site: Other

Number of metastatic organs (5 categories)

Presence or absence of clinically important comorbidities

Presence or absence of clinically important concomitant drugs

Less than 1 year from diagnosis to the initiation of systemic therapy

Karnofsky Performance Status < 80%

Hemoglobin value below the lower normal limit

Corrected calcium value above the upper normal limit

Neutrophil count above the upper normal limit

Platelet count above the upper normal limit

IMDC risk group

Number of risk factors (7 categories)

Breakdown of IMDC risk factors by the number of risk factors

Summary statistics will be calculated for continuous variables.

Analysis content

The following aggregation will be performed for endpoints:

A frequency table (number of cases, percentage (%)) will be created

for categorical variables.

A frequency table (number of cases, percentage (%)) will also be created for details regarding clinically important comorbidities and

concomitant drugs

### [Division of categorical variables]

| Factor | Category |
|---|---|
| Age (2 categories) | <75 years; ≥75 years |
| Age (3 categories) | <65 years; ≥65 years and <75 years; ≥75 years |
| Gender | Male; Female |
| Body mass index (3categories) | $<25 \text{ kg/m}^2$ ; $\ge 25 \text{ kg/m}^2$ ; Unknown |
| C-reactive protein (3 categories) | <5 mg/L; ≥5 mg/L; Unknown |
| Estimated glomerular filtration rate | <60; ≥60; Unknown |
| (3 categories) | |
| Smoking history | No (no past smoking); No (history of past |
| | smoking); Yes; Unknown |

**ECOG Performance Status** 0; 1; 2; 3; 4 ECOG Performance Status (1) 0: 1: >2ECOG Performance Status (2) 0 or 1; >2TX: T0; T1; T1a; T1b; T2; T2a; T2b; T3; T3a; Invasion depth (T factor) T3b; T3c; T4; Unknown Lymph node metastasis (N factor) NX: N0: N1: Unknown Distant metastasis (M factor) MX; M0; M1; Unknown Tumor histological type Clear cell renal cell carcinoma; Papillary renal cell carcinoma; Chromophobe renal cell carcinoma; Other Presence or absence of sarcomatoid No: Yes component Fuhrman grade Grade 1; Grade 2; Grade 3; Grade 4; Unknown Grade 1 or Grade 2: Grade 3 or Grade 4: Fuhrman grade (3 categories) Unknown -; ±; 1+; 2+; 3+; Not measured Proteinuria Performance of nephrectomy No: Yes: Unknown Presence or absence of metastasis No: Yes: Unknown Metastatic site Lung; Liver; Bone; Brain; Regional lymph node; Distant lymph node; Other No; Yes; Unknown Metastatic site: Lung Metastatic site: Liver No; Yes; Unknown Metastatic site: Bone No; Yes; Unknown No; Yes; Unknown Metastatic site: Brain Metastatic site: Regional lymph No: Yes: Unknown node Metastatic site: Distant lymph node No: Yes: Unknown Metastatic site: Other No: Yes: Unknown Number of metastatic organs 0; 1; 2; 3; >4No: Yes: Unknown Presence or absence of clinically important comorbidities Presence or absence of clinically No: Yes: Unknown important concomitant drugs Yes; No Less than 1 year from diagnosis to the initiation of systemic therapy Karnofsky Performance Status Yes: No <80% Hemoglobin value below the lower Yes; No normal limit Corrected calcium value above the Yes: No upper normal limit

| Neutrophil count above the upper | Yes; No |
|----------------------------------|----------------------------------|
| normal limit | |
| Platelet count above the upper | Yes/; No |
| normal limit | |
| IMDC risk group | Low risk; Medium risk; High risk |
| Number of risk factors (7 | 0; 1; 2; 3; 4; 5; 6 |
| categories) | |

# Analysis of secondary objectives

# 7.2.2.2 Real-world progression-free survival

Source

Efficacy analysis set

population Endpoint

Real-world PFS

Analysis content

For the endpoint, the median and its 95% confidence interval will be calculated using the Kaplan–Meier method. In addition, the Kaplan–Meier curve will be plotted, and the PFS rate for every 12 months and its 95% confidence interval will be calculated. Greenwood's formula will be used to calculate the confidence interval for the PFS rate. In addition, the number of event-onset cases and the number of censored cases will be presented. A frequency table (number of cases, percentage (%)) will be created, considering the reasons for the event and reasons for censoring.

In order to evaluate the observation period, the median observation period and its 95% confidence interval will be calculated by estimating the reverse Kaplan-Meier curve in which censoring patients are regarded as patients with events and patients with events

are regarded as censoring patients.

#### [Division of categorical variables]

| Bivision of categorical variables | |
|---|---|
| Factor | Category |
| Reasons for the event | Disease progression after the start of avelumab plus axitinib; Death |
| Reasons for the censoring | No disease progression during or after first-line therapy; second-line therapy started; nephrectomy performed |

### 7.2.2.3 Overall survival (OS)

Source . Efficacy analysis set

population

content

Efficacy analysis se

Endpoint : OS

Analysis . Fo

For the endpoint, the median and its 95% confidence interval will be calculated using the Kaplan–Meier method. In addition, the Kaplan–Meier curve will be plotted, and the survival rate for every 12 months

#### PFIZER CONFIDENTIAL

CT24-WI-GL03-RF03 2.0 Non-Interventional Statistical Analysis Plan For Secondary Data Collection Study 01-Jun-2020 

and its 95% confidence interval will be calculated. Greenwood's formula will be used to calculate the confidence interval for the survival rate.

In addition, a frequency table (number of cases, percentage (%)) will be created, considering the event onset, censoring, reasons for the event, and reasons for censoring.

In order to evaluate the observation period, the median observation period and its 95% confidence interval will be calculated by estimating the reverse Kaplan-Meier curve in which censoring patients are regarded as patients with events and patients with events are regarded as censoring patients.

#### [Division of categorical variables]

| Factor | Category |
|---|---|
| Reasons for the event (cause of | Death from primary disease; Death related to |
| death) | avelumab plus axitinib combination therapy; |
| , | Death not related to avelumab plus axitinib |
| | combination therapy |
| Reasons for censoring | Survival; Untraceable |

# 7.2.2.4 Objective response rate (ORR)

Source population

Efficacy analysis set

**Endpoints** 

ORR

Presence or absence of confirmation of BOR to treatment

Evaluation method

Determination of BOR (tumor assessment)

Analysis content The number of target cases, number of objective responding cases, and objective response rate and its 95% confidence interval will be

calculated to establish the ORR of the endpoint.

In addition, the Clopper–Pearson method will be used to calculate the

confidence interval.

In addition, a frequency table (number of cases, percentage (%)) will also be created, considering the achievement of BOR to treatment, evaluation method, and determination of BOR (tumor assessment).

#### [Division of categorical variables]

| <u>- </u> | |
|-----------------------------------------------|---------------------------|
| Factor | Category |
| Objective response to avelumab | Objective response |
| plus axitinib combination therapy | |
| Achievement of the best overall | No; Yes |
| response to treatment | |
| Evaluation method | RECIST; Other than RECIST |

| Determination of best overall | CR; PR; SD; PD; NE |
|-------------------------------|--------------------|
| response (tumor assessment) | |

CR, complete response; PR, partial response; PD, progressive disease; NE, not evaluable for response.

# 7.2.2.5 Best overall response for primary lesions

Source

population

Efficacy analysis set

**Endpoints** ORR

Presence or absence of confirmation of BOR to treatment

Evaluation method

Determination of BOR (tumor assessment)

Analysis content The number of target cases, number of objective responding cases, and objective response rate and its 95% confidence interval will be

calculated to establish the ORR of the endpoint.

In addition, the Clopper–Pearson method will be used to calculate the

confidence interval.

A frequency table (number of cases, percentage (%]) will also be created, considering the achievement of BOR to treatment, evaluation

method, and determination of BOR (tumor assessment).

# [Division of categorical variables]

| Factor | Category |
|-------------------------------|---------------------------|
| Objective response of primary | Objective response |
| lesions | |
| Achievement of best overall | No; Yes |
| response to treatment | |
| Evaluation method | RECIST; Other than RECIST |
| Determination of best overall | CR; PR; SD; PD; NE |
| response (tumor assessment) | |

CR, complete response; PR, partial response; PD, progressive disease; NE, not evaluable for response.

# 7.2.2.6 Time to treatment discontinuation (TTD) of avelumab plus axitinib combination therapy as first-line therapy

Efficacy analysis set Source

population Endpoints

TTD of avelumab plus axitinib combination therapy as first-line

therapy

TTD of avelumab as first-line therapy TTD of axitinib as first-line therapy

Analysis content Considering the endpoints, the median and its 95% confidence interval will be calculated using the Kaplan-Meier method. In addition, the Kaplan-Meier curve will be plotted, and the survival

#### PFIZER CONFIDENTIAL

CT24-WI-GL03-RF03 2.0 Non-Interventional Statistical Analysis Plan For Secondary Data Collection Study 01-Jun-2020 

rate for every 3 months, along with its 95% confidence interval, will be calculated. Greenwood's formula will be used to calculate the confidence interval for the survival rate.

In addition, a frequency table (number of cases, percentage (%)])will be created, considering the event onset, censoring, reasons for the event, and reasons for censoring.

# [Division of categorical variables]

| Factor | Category |
|---------------------------|-------------------------------------------|
| Reasons for the event | Disease progression/adverse event/other |
| | (death)/other (excluding death) |
| Reasons for the censoring | Treatment ongoing; Discontinuation due to |
| | efficacy |

# 7.2.2.7 Treatment patterns for avelumab plus axitinib combination therapy as first-line therapy in a real-world setting

Source:

FAS, Efficacy analysis set

population

Endpoints : Continuous variables

Duration of treatment for avelumab plus axitinib (days)

Duration of treatment for avelumab (days) Duration of treatment for axitinib (days) Initial dose of avelumab [daily dose (mg)] Initial dose of axitinib [daily dose (mg)]

Avelumab dose intensity (DI)

Axitinib DI

Axitinib relative DI (RDI)<sup>1)</sup>

#### Categorical variables

Initial dose of avelumab [daily dose (mg)]

Initial dose of axitinib [daily dose (mg)]

Presence or absence of changes in the avelumab dose <sup>2)</sup>

Presence or absence of changes in the avelumab dose (dose

reduction)<sup>2)</sup>

Reason for changes in the avelumab dose (dose reduction) <sup>2)3)</sup>

Presence or absence of change in the avelumab dose (dose increase)

2)

Termination of avelumab administration

Reason for termination of avelumab administration

Presence or absence of changes in the axitinib dose 2)

Presence or absence of changes in the axitinib dose (dose reduction)

Reason for change in the dose of axitinib (dose reduction) <sup>2)3)</sup>

Presence or absence of changes in the axitinib dose (dose increase) 2)

Termination of axitinib administration

#### Reason for termination of axitinib administration

#### Notes:

- 1) 10 mg/day is set as the criterion.
- 2) Dose changes will be aggregated based on the input items, considering the administration status in the case report form. The criteria for dose changes will be determined based on the record of the immediately preceding administration for both avelumab and axitinib.
- 3) Considering the reason for dose reduction, if the same reason is documented in multiple records of the case, each reason will be counted as one case.

# Analysis content

The following aggregation will be performed for the endpoints:

Summary statistics will be calculated for continuous variables.

A frequency table (number of cases, percentage (%]) will be created for categorical variables.

In addition, a list presenting the reasons underlying the changes in the avelumab dose (dose increase) and those underlying changes in the axitinib dose (dose increase) will be created.

Furthermore, a swimmer plot with the date of initiation as the avelumab + axitinib administration start date (earlier date if they are different) will be created.

# [Division of categorical variables]

| Factor | Category |
|---|---|
| Initial avelumab dose [daily dose | <10 mg/kg; 10 mg/kg; >10 mg/kg |
| (mg)] | |
| Initial axitinib dose [daily dose (mg)] | $<2$ mg; $\geq$ 2 mg and $<$ 5 mg; $\geq$ 5 mg and $<$ 10 mg; |
| | <10 mg; 10 mg; >10 mg |
| Presence or absence of changes in the | No; Yes |
| avelumab dose | |
| Presence or absence of changes in the | No; Yes |
| avelumab dose (dose reduction) | |
| Reason for changes in the avelumab | Disease progression; Adverse event; |
| dose (dose reduction) | discontinuation due to efficacy; Other |
| Presence or absence of changes in the | No; Yes |
| avelumab dose (dose increase) | |
| Termination of avelumab | No; Yes |
| administration | |
| Reason for termination of avelumab | Disease progression; Adverse event; |
| administration | discontinuation due to efficacy; Other |
| Presence or absence of changes in the | No; Yes |
| axitinib dose | |

| Presence or absence of changes in the | No; Yes |
|---|---|
| axitinib dose (dose reduction) | |
| Reason for changes in the axitinib | Disease progression; Adverse event; |
| dose (dose reduction) | discontinuation due to efficacy; Other |
| Presence or absence of changes in the | No; Yes |
| axitinib dose (dose increase) | |
| Termination of axitinib administration | No; Yes |
| Reason for termination of axitinib | Disease progression; Adverse event; |
| administration | discontinuation due to efficacy; Other |

# 7.2.2.8 Clinical use of corticosteroids for immune-related adverse events (irAEs) occurring during the course of avelumab plus axitinib combination therapy

Source

FAS, Efficacy analysis set

population Endpoints

Continuous variable

Duration of treatment for corticosteroids (days)

Categorical variables

Administration of corticosteroid therapy for irAEs

Administration of high-dose corticosteroid therapy for irAEs

(prednisolone-equivalent of ≥40 mg)

Analysis content

The following aggregation will be performed for the endpoints: Summary statistics will be calculated for continuous variables.

A frequency table (number of cases, percentage (%)) will be created

for categorical variables.

In addition, a frequency table (number of cases, percentage (%)) will

also be created for the details of other drugs.

#### [Division of categorical variables]

| Factor | Category |
|----------------------------------|------------------|
| Administration of corticosteroid | No; Yes; Unknown |
| therapy for irAEs | |
| Administration of high-dose | No; Yes |
| corticosteroid therapy for irAEs | |

irAEs, immune-related adverse events

# 7.2.2.9 Pre-treatment and treatment of infusion-related reactions caused by avelumab

Source

FAS, Efficacy analysis set

population Endpoints

· Presence or absence of premedication

Detailed name of the drug

Presence or absence of treatment and coping

Analysis: A frequency table (number of cases, percentage (%)) will be created

c o n t e n t for the endpoints.

# [Division of categorical variables]

| Factor | Category |
|----------------------------------|------------------|
| Presence or absence of | No; Yes; Unknown |
| premedication | |
| Presence or absence of treatment | No; Yes; Unknown |
| and coping | |

# 7.2.2.10 Subsequent treatment of avelumab plus axitinib combination therapy

Source: FAS, Efficacy analysis set

population

Endpoints · Continuous variables

Second-line therapy period (days)

The period from the end date of first-line therapy to the beginning of

second-line therapy (days)

Categorical variables

Performance of nephrectomy after avelumab plus axitinib

combination therapy

Presence or absence of second-line therapy

Drug category

Second-line therapy regimen by drug category

Analysis: The content Sum

The following aggregation will be performed for the endpoints: Summary statistics will be calculated for continuous variables.

The period from the end date of first-line therapy to the beginning of second-line therapy (days) will also be estimated, considering the

reason for termination of administration.

A frequency table (number of cases, percentage (%)) will be created

for categorical variables.

# [Division of categorical variables]

| Factor | Category |
|------------------------------------|----------------------|
| Performance of nephrectomy after | No; Yes |
| avelumab plus axitinib combination | |
| therapy | |
| Presence or absence of second-line | No; Yes; Unknown |
| therapy | |
| Drug category | TKI; mTOR; IO; Other |

mTOR, mammalian target of rapamycin; IO, immunotherapy; TKI, tyrosine kinase inhibitor.

| <br> |
|------|

| CCI |
|-----|

#### 8 LIST OF TABLES AND TABLE SHELLS

Not applicable

#### 9 REFERENCES

Not applicable

#### 10 APPENDIXES

Not applicable

#### 10.1 APPENDIX 1: DATA DERIVATION DETAILS

Not applicable

# A1.1 Definition and use of visit windows in reporting

Not applicable

# A1.2 Further definition of endpoints

Not applicable

# 10.2 APPENDIX 2: ADDITIONAL STATISTICAL METHODOLOGY DETAILS

Not applicable

# A2.1 Further details regarding the statistical methods

Not applicable

# 10.3 APPENDIX 3: DIAGNOSIS AND PROCEDURE CODES USED IN THE STUDY

Not applicable